CLINICAL TRIAL: NCT04567771
Title: A Comparison of Acute Toxicities Between Patients Treated With Protons or Intensity-Modulated Radiation Therapy for Post-Operative Treatment of Endometrial or Cervical Cancers
Brief Title: Comparison of Proton or Intensity Modulated Radiation Therapy After Surgery for Endometrial or Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1961; NCI-2020-06936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ROR1904 (Other: Mayo Clinic Radiation Oncology); 19-004792 (Other: Mayo Clinic Institutional Review Board); MC1961 (Other: Mayo Clinic); NCT04745650 (obsolete NCT alias)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervical Carcinoma; Endometrial Carcinoma; Endometriosis; Pelvic Inflammatory Disease
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Endometriosis; Pelvic Inflammatory Disease | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (radiation therapy, questionnaires) (Experimental): Patients undergo standard of care proton or intensity modulated radiation therapy. Patients also complete quality of life questionnaires and adverse event assessments over 10-15 minutes each at baseline, at the end of radiation therapy, and at 1 month, 1 year, and 3 years post-radiation therapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete quality of life questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete adverse event assessments
Radiation: Radiation Therapy — Undergo proton or intensity modulated radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This early phase I trial compares the side effects between patients treated with proton radiation therapy versus intensity modulated radiation therapy after surgery for the treatment of endometrial or cervical cancer. Radiation therapy uses high energy protons or x-rays to kill tumor cells and shrink tumors. Using quality of life questionnaires and adverse event assessments may help doctors learn whether proton radiation therapy is associated with lower acute gastrointestinal toxicities at the end of treatment compared to intensity modulated radiation therapy in patients with endometrial or cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether proton radiation therapy (RT) is associated with lower acute gastrointestinal toxicities at the end of treatment compared to intensity modulated radiation therapy (IMRT) as measured with the Expanded Prostate Cancer Index Composite (EPIC) bowel domain.

SECONDARY OBJECTIVES:

I. To examine the association of bowel and bladder dose-volume histogram (DVH) with bowel and bladder toxicities, respectively.

II. To assess whether urinary toxicity rate is improved with proton RT compared to IMRT as measured with the EPIC urinary domain.

III. To determine if well-being is improved with proton RT compared to IMRT as measured by the Functional Assessment of Cancer Therapy (FACT) cervix domain.

IV. To determine if proton RT reduces grade 2+ hematologic toxicities (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.0) compared to IMRT.

V. Evaluate progression-free and overall survival between patients receiving proton RT and IMRT.

VI. To determine if proton RT improves overall patient quality of life compared to IMRT using the European Quality of Life Five Dimension (EQ-5D) questionnaire.

EXPLORATORY OBJECTIVES:

I. Evaluate ability to tolerate chemotherapy concurrent or after RT. II. Correlate bone marrow DVH with blood marrow function, and ability to tolerate chemotherapy concurrently or after RT.

III. Correlate bowel and skin DVH with acute toxicity. IV. To evaluate patient-reported gastrointestinal (GI) toxicities as a predictor of assigned treatment regimen, as well as physician-reported GI toxicities as a predictor of assigned treatment regimen.

V. Confirm the validity of the EPIC bowel and urinary domains when referencing the last 7 days.

OUTLINE:

Patients undergo standard of care proton or intensity modulated radiation therapy. Patients also complete quality of life questionnaires and adverse event assessments over 10-15 minutes each at baseline, at the end of radiation therapy, and at 1 month, 1 year, and 3 years post-radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of cervical or endometrial cancer
* Must have undergone an open or robotic hysterectomy (total abdominal, vaginal, radical, or total laparoscopic) for carcinoma of the cervix or endometrium
* History and physical prior to registration
* Documentation of history of:

  * Smoking status
  * Pelvic infection
  * Pelvic inflammatory disease
  * Endometriosis
* Planned to receive either proton or IMRT radiation treatment, with use of rectal balloon, at any Mayo Clinic site
* Plan for RT to pelvis with or without para-aortic lymph node irradiation
* If received high-dose chemotherapy prior to registration, last dose must have been given >= 21 days prior to start of RT
* Complete blood count (CBC) performed within 21 days prior to registration
* Computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET)/CT, or PET/MRI for staging before registration; may be pre-operative (op) or post-op
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Provide written informed consent
* Willing to complete quality of life (QOL) questionnaires

Exclusion Criteria:

* Receiving external beam boost dose during RT
* Distant metastases
* Gross disease at time of RT
* Histology of endometrial stromal sarcoma, leiomyosarcoma, melanoma or small cell carcinomas
* Patients who exceed the weight/size limits of the treatment table
* Positive or close surgical margins (=< 3 mm)
* Prior RT to the pelvis
* Planned to receive inguinal node RT
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be immunosuppressive.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Other major medical illness which requires hospitalization or precludes study therapy at the time of registration
* Patients unwilling to have rectal balloon placed on a daily basis during RT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Prostate Cancer Index Composite (EPIC) Bowel score | Baseline up to 3 years post-radiation therapy (RT)
  Will be examined using analysis of covariance.

SECONDARY OUTCOMES:
Bowel and bladder dose-volume histogram (DVH) parameters | Up to 3 years post-RT
  Will be examined in association with the change in EPIC Bowel and Urinary scores using analysis of covariance, considering the DVH variables as model covariates.
Change in EPIC Urinary score | Baseline up to 5 weeks
  Will be examined using analysis of covariance.
Well-being | Up to 3 years post-RT
  Measured by the Functional Assessment of Cancer Therapy cervix domain. Will be examined using analysis of covariance.
Incidence of grade 2+ hematologic toxicities | Up to 3 years post-RT
  Measured by Common Terminology Criteria for Adverse Events version 4.0. Will be examined using logistic regression.
Progression-free survival | Up to 3 years post-RT
  Will be examined using survival methods. Cumulative probability of progression rates will be calculated treating death as a competing risk. Cox models will be used to assess the association of treatment received (proton RT versus intensity modulated radiation therapy [IMRT]).
Overall survival (OS) | Up to 3 years post-RT
  Will be examined using survival methods. Estimates of OS will be calculated using the Kaplan Meier method. Cox models will be used to assess the association of treatment received (proton RT versus IMRT).
Change in overall patient quality of life | Baseline up to 3 years post-RT
  Measured by the European Quality of Life Five Dimension Five Level Scale Questionnaire. Will be examined using analysis of covariance.

CONTACTS AND LOCATIONS:
Overall Officials: Allison E. Garda, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials